CLINICAL TRIAL: NCT01803126
Title: A Proposed Study of Atherosclerotic Plaques in Leg Arteries
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Sponsor
Other Study IDs: 56-RW-024
Record Dates: First submitted 2012-09-18; First posted 2013-03-04 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Vascular Disease; Diabetes
Keywords: atherosclerosis
MeSH Terms: conditions — Vascular Diseases; Diabetes Mellitus; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- atherosclerosis: No treatment.

SUMMARY:
Biofilm has been identified as the major bacterial phenotype contributing to atherosclerosis. It has become very important to evaluate atherosclerosis and the role of biofilm using advanced technologies. It is also important to understand wound biofilm at a genetic and a molecular level.

DETAILED DESCRIPTION:
High throughput pyrosequencing is opening new doors in nucleic acid analysis. 454 Roche has developed sequencing instrumentation which has the ability to sequence not only genomic DNA (gDNA) but also derivatives of messenger RNA (mRNA) and 16s ribosomal DNA (rDNA). This technology has the potential to survey the nucleic acids involved within a mixed population of species, such as atherosclerotic biofilm. In addition to transcriptome science; proteome, metabolome, and other -omic sciences are advancing rapidly. Examining atherosclerotic plaque using transcriptome, proteome, metabolome, and other -omic approaches may provide valuable insight into the wound's microecology.

ELIGIBILITY:
Inclusion Criteria:

1. The subject with identifying leg or legs that were amputated for vascular disease and/or diabetes.
2. The subject must be 18 years of age or older.

Exclusion Criteria:

* The subject will be excluded if they have had a traumatic amputation which did not involve vascular disease and/or diabetes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject with vascular disease or diabetes.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
To study the role of biofilm in the hardening of the arteries. The study will evaluate the hardening of the arteries found in legs that have been amputated because of vascular disease and/or diabetes. | 1 year
  Amputated legs will be dissected and en bloc removal of atherosclerotic arteries will be performed within the pathology department of TTUHSC. Preferred artery specimen will be grossly involved arteries that are 5-10 cm in length. The specimens would be flash frozen and stored at -81 degrees within the department until analysis could be undertaken. Frozen tissue would be transferred to the site for further testing (R&T) once the accrual goal was met. This technology has the potential to survey the nucleic acids involved within a mixed population of species, such as atherosclerotic biofilm. In addition to transcriptome science; proteome, metabolome, and other -omic sciences are advancing rapidly. Examining atherosclerotic plaque using transcriptome, proteome, metabolome, and other -omic approaches may provide valuable insight into the wound's microecology.

CONTACTS AND LOCATIONS:
Overall Officials: Randall D Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No